CLINICAL TRIAL: NCT00253994
Title: Auricular Acupuncture in the Treatment of Acute Pain Syndromes (AATAPS) Pilot
Brief Title: Auricular Acupuncture for Acute Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: MIL-03-01; MGMC IRB #: FMG20030009H
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
* Auricular Acupuncture in the Treatment of Acute Pain Syndromes (AATAPS)
* Study Period: August 1, 2003 - December 31, 2004

DETAILED DESCRIPTION:
Although inroads in the study of acupuncture for acute pain conditions have been made, there are still critical gaps in the literature in both basic/mechanistic and clinical areas. Very little is know about what impact conservative, easily transportable and administered treatments, such as acupuncture, might have in preserving military battlefield readiness. The proposed research proposal is an incremental step with the ultimate goal to increase the knowledge base and expand clinical applications of acupuncture for acute pain conditions that are relevant to military personnel and operations.The purpose of this proposal is to conduct a scientifically rigorous investigation of auricular acupuncture for the treatment of acute pain in the emergency room setting at a military hospital using a two phase clinical trial design. This pragmatic investigation will provide a unique opportunity to develop clinically relevant questions that can be further evaluated in the context of basic science and more robust clinical trial designs. The specific aims of this study are to 1) Determine the feasibility of conducting a clinical trial of auricular acupuncture in the treatment of military personnel with acute pain who present to the emergency room at Andrews Air Force Base, using a pilot two phase clinical trial approach and 2) Gather data on the effect size of auricular acupuncture in treating acute pain conditions. Persons presenting to the emergency room at Malcolm Grow with acute pain syndromes that do not require medical attention beyond pain management strategies will be invited to participate in the study and asked for informed consent. The study will involve a preliminary pilot test period during which 20 persons are entered into a consecutive case series study to test the feasibility of collecting data and implementing the treatment procedures in the busy emergency room setting. Treatment will involve auricular acupuncture using SEDATELEC Aiguille Semi-Permanent (ASP) needles bilaterally at two acupuncture points - Cingulate Gyrus and Thalamic Nuclei. Baseline demographic and pain indicator information will be collected prior to treatment. Follow-up data on pain levels and medication use will occur prior to leaving the ER and 24 hours following treatment. The primary endpoint is change in pain levels at 24 hours, as measured by the verbal Numerical Rating Scale (NRS). 24 hour follow-up will occur via the telephone. Following successful completion of the preliminary study, a two arm, randomized clinical pilot trial of 100 participants (N = 50 per arm) will be conducted using the same protocol as the case series study. Patients will be randomized to either usual emergency medical care or acupuncture + medical co-management. Follow-up data will be collected on the schedule outlined above by assessors blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pain syndrome
* Written Informed Consent
* Over the age of 18

Exclusion Criteria:

* Unwilling or unable to participate in study treatment and follow-up
* Require medical intervention other than pain management
* Pregnant or nursing
* Unable to give informed consent for any reason
* Extreme pain
* Allergic reaction to adhesive tape, gold or other components of the acupuncture needles
* Admitted to the hospital for care

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-08; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was current level of pain, as measured by the verbal Numerical Rating Scale (NRS | Before leaving the ER; 24 hours post-treatment

SECONDARY OUTCOMES:
Change in Medication Use, if any | Baseline; 24 hours post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Goertz, DC, PhD, Principal Investigator — Samueli Institute for Information Biology
Locations (1):
- Malcolm Grow Medical Center, Andrews Air Force Base, Andrews Air Force Base Census Designated Place, Maryland, United States